CLINICAL TRIAL: NCT00794378
Title: A Single-Center, Pediatric, Comparative Taste Test of Desloratadine and Cetirizine Antihistamine Syrup Medications
Brief Title: Taste Test Between Desloratadine and Cetirizine Syrup in Children (Study P03829)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: P03829
Expanded Access: Available
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — desloratadine; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Desloratadine and Cetirizine Crossover (Experimental): To compare the preference in taste between desloratadine and cetirizine.
  Interventions: Drug: Desloratadine (Clarinex); Drug: Cetirizine (Zyrtec)

INTERVENTIONS:
Drug: Desloratadine (Clarinex) — Each subject received 5 mL of desloratadine syrup one time
  Other Names: SCH 034117, Clarinex
Drug: Cetirizine (Zyrtec) — Each subject received 5 mL of cetirizine syrup
  Other Names: Zyrtec

SUMMARY:
This study was conducted to compare the taste acceptability of Zyrtec syrup with desloratadine syrup in children. Children between 6 and 11 years of age received 5 mL of each syrup, separated by 15 to 20 minutes on a single day.

DETAILED DESCRIPTION:
This study is a cross-over study design.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be:

* Between 6 and 11 years of age in good general health
* Premenarcheal if female

Exclusion Criteria:

Subjects who:

* Have known allergies or sensitivities to either of the drug formulations
* Have a medical condition that may interfere with the subject's ability to discriminate between tastes
* Have used any antihistamines within 24 hours prior to dosing
* Were taking sedatives, tranquilizers, or monoamine oxidase inhibitor drugs
* Were involved in another clinical or market research study within the past 30 days

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2004-11; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Taste acceptability as determined from smiley-face scale of 1 (frowning child) to 5 (happy child face). | During the only study visit

SECONDARY OUTCOMES:
Taste flavor preference between bubble-gum, banana-grape, or grape flavors | During the only study visit
Adverse Events | During the only study visit